CLINICAL TRIAL: NCT01848418
Title: Conception of an ICF Core Set for Systemic Sclerosis
Acronym: SCISCIF
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Cabinet d'étude INTERLIS (Unknown); Ecole des Hautes Etudes en Santé Publique (Other); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: AOR - 10050
Record Dates: First submitted 2013-05-03; First posted 2013-05-07 (Estimated); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Systemic Sclerosis
Keywords: ICF; Core sets; Systemic sclerosis; Function; Evaluation
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to create and validate an ICF core Set for Systemic sclerosis

DETAILED DESCRIPTION:
In 2002 was published WHO's International Classification of Functioning, Disability and Health (ICF). ICF defines disability as "the negative aspects of the interaction between an individual (with a health condition) and that individual's contextual factors (personal and environmental factors)". Interactions are specified in five domains, classified from body, individual and societal perspectives by means of two lists: a list of body functions and structure, and a list of domains of activity and participation. Since an individual's functioning and disability occurs in a context, the ICF also includes a list of environmental factors.

ICF core sets, which are short lists of ICF categories relevant for specific conditions, serve as practical tools for clinical practice and allow standardisation of data for health information and research. Core sets have already been developed and validated for several musculoskeletal diseases, such as low back pain, osteoarthritis, or osteoporosis, but not yet for systemic sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 and older
* Diagnosis of ScS made according to ACR and/or Leroy et Medsger criteria
* Patient giving his informed consent to participate in the study

Exclusion Criteria:

* Severe chronic disease associated with ScS : stroke, multiple sclerosis, Parkinson's disease,…
* Cognitive or behavioral disorders making assessment impossible
* Inability to speak and write French

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female aged 18 and older with a diagnosis of ScS made according to ACR and/or Leroy et Medsger criteria
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2012-10-27 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Validation of an ICF core Set for Systemic sclerosis | Between the 13th and 24th month
  Submit the list of items to a cohort of 100 patients and experts.

SECONDARY OUTCOMES:
Translation of concepts identified such as items ICF (linking). | Between the 10th and 12th month
  Translation of extracted data and set up the core set
Creation of a database from a qualitative survey | During the first 9 months
  This database will be elaborated considering information from a qualitative survey of 100 patients, a consultation with experts and a review of the literature

CONTACTS AND LOCATIONS:
Overall Officials: Agathe Papelard, MD, Principal Investigator — Cochin Hospital
Locations (1):
- Cochin Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cieza A, Geyh S, Chatterji S, Kostanjsek N, Ustun B, Stucki G. ICF linking rules: an update based on lessons learned. J Rehabil Med. 2005 Jul;37(4):212-8. doi: 10.1080/16501970510040263. PMID 16024476
- [Background] Cieza A, Geyh S, Chatterji S, Kostanjsek N, Ustun BT, Stucki G. Identification of candidate categories of the International Classification of Functioning Disability and Health (ICF) for a Generic ICF Core Set based on regression modelling. BMC Med Res Methodol. 2006 Jul 27;6:36. doi: 10.1186/1471-2288-6-36. PMID 16872536
- [Background] Clements PJ. Systemic sclerosis (scleroderma) and related disorders: clinical aspects. Baillieres Best Pract Res Clin Rheumatol. 2000 Mar;14(1):1-16. doi: 10.1053/berh.1999.0074. PMID 10882211
- [Background] Coenen M, Cieza A, Stamm TA, Amann E, Kollerits B, Stucki G. Validation of the International Classification of Functioning, Disability and Health (ICF) Core Set for rheumatoid arthritis from the patient perspective using focus groups. Arthritis Res Ther. 2006;8(4):R84. doi: 10.1186/ar1956. PMID 16684371
- [Result] Daste C, Abdoul H, Foissac F, Papelard A, Alami S, Kwakkenbos L, Carrier ME, Lefevre-Colau MM, Thombs BD, Poiraudeau S, Rannou F, Mouthon L, Nguyen C. Development of a new patient-reported outcome measure to assess activities and participation in people with systemic sclerosis: the Cochin 17-item Scleroderma Functional scale. Br J Dermatol. 2020 Oct;183(4):710-718. doi: 10.1111/bjd.18922. Epub 2020 Mar 18. PMID 32017013
- [Derived] Papelard A, Daste C, Alami S, Sanchez K, Roren A, Segretin F, Lefevre-Colau MM, Rannou F, Mouthon L, Poiraudeau S, Nguyen C. Construction of an ICF core set and ICF-based questionnaire assessing activities and participation in patients with systemic sclerosis. Rheumatology (Oxford). 2019 Dec 1;58(12):2260-2272. doi: 10.1093/rheumatology/kez209. PMID 31219594